CLINICAL TRIAL: NCT05812924
Title: A Novel Therapy for Breast Cancer Survivors With Genitourinary Syndrome of Menopause
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kristin E. Rojas, MD, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20221120
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platelet-rich plasma (PRP) Group (Experimental): Participants will undergo two sessions of platelet-rich plasma (PRP) injections to the vulva/vagina one month apart.
  Interventions: Biological: Platelet-rich plasma (PRP)

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP) — 0.1-0.2 mL injections of platelet-rich plasma (PRP) will be injected to the vulvovaginal area. The injections will be placed every 5mm and at an angle of 60° into the mucosa and lamina propria of the posterior wall of the vagina.

SUMMARY:
The purpose of this study is to determine whether platelet rich plasma (PRP) injections to the vulva and vagina will improve symptoms of genitourinary syndrome of menopause (GSM) in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are age 18 years and older
* Patients must have a history of biopsy-proven Ductal carcinoma in situ (DCIS) or Stage I-III breast cancer and must be currently undergoing treatment or have completed primary treatment.
* Patients must be found to have a vaginal health index (VHI) score of <15.
* Patients may be currently using endocrine therapy (ovarian function suppression, tamoxifen, or aromatase inhibitors). Patients not currently using endocrine therapy will also be eligible for participation since patients more than 5 or 10 years from diagnosis (and therefore having completed adjuvant endocrine therapy) may be enrolled.
* Some patients with triple negative breast cancer who receive chemotherapy also experience GSM related to ovarian function decline outside of the setting of ovarian suppression, and therefore patients with either ER+ or ER- breast cancer will be allowed to participate.
* Patients must provide written informed consent for participation in this study.
* Patients are allowed to have used non-hormonal moisturizers but if they have previously used hormonal moisturizers, they will be asked to stop the use for one month prior to the first planned treatment, termed the "washout period", if needed.

Exclusion Criteria:

* Patients with any systemic or topical hormone replacement therapy within 3 months prior to enrollment, known genital infection, coagulation disorders, or on anticoagulant therapy or turmeric-containing supplements within the prior 2 weeks will be excluded.
* Women who are pregnant or who plan to become pregnant within the following six months will be excluded since the impact of recent PRP injections to the vulva and the impact on obstetric injury during vaginal delivery has not been studied.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in GSM symptoms as measured by vulvovaginal symptom questionnaire (VSQ). | Baseline, up to 31 weeks
  The VSQ is a 21-question survey that specifically asks about GSM symptoms and their impact on quality of life and sexual function. Vaginal and vulvar symptoms will be self-reported using validated VSQ modified to 4-point Likert scores. VSQ consists of a series of questions, each of which is rated as 0 (never), 1(rarely), 2(sometimes), 3 (frequently). Lower scores indicate better health. Each question is analyzed separately; there is no overall score reported.

SECONDARY OUTCOMES:
Change in Vaginal health index (VHI) Score | Baseline, up to 31 weeks
  VHI assesses post menopausal symptoms such as dryness, burning, and irritation. Each component is scored on a scale of 1 (worst) to 5 (best). Lower scores indicate more severe atrophy.
Change in validated female sexual function index (FSFI) | Baseline, up to 31 weeks
  Change in validated female sexual function index (FSFI) is determined by the participant response to the female sexual function index (FSFI) questionnaire. The FSFI is a questionnaire competed by the participant and is designed to measure sexual functioning by assessing six areas of sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. Scores range from 2 to 36. Higher scores indicate better sexual function.
Change in sexual-related distress (FSDS-R). | Baseline, up to 31 weeks
  Change in validated female sexual distress is determined by participant response to the female sexual distress survey-revised (FSDS-R). The FSDS-R is a self reported questionnaire that asks participants to rate distress related to low sexual desire. Responses to the items on the Likert-type scale consist of never (0), rarely (1), sometimes (2), often (3), or always (4). The lowest score that can be obtained from the FSDS-R is "0" and the highest score is "52". Higher scores indicate higher levels of sexual distress.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Rojas, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No